CLINICAL TRIAL: NCT01217580
Title: Analgesic Efficacy of Ultrasound Guided Transversus Abdominis Plane Block After Cesarean Delivery in Patients With a BMI > 30
Brief Title: Pain Relief Study of Ultrasound Guided Transverse Abdominis Plane(TAP)Block
Acronym: TAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not feasible to perform at one institution with the amount of subjects that were needed to complete it.
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Stuart Hart, Director of Obstetric Anesthesiology, Ochsner Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010.091.C; PI-Hart (Other: Ochnser Clinic Foundation Institutional Review Board)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Cesarean Section
Keywords: c-section; cesarean section; TAP block; pain; pain after delivery; pain after C-section; pain after C-section delivery; pain after cesarean delivery; pain after cesarean
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20 ml per side of 0.5% ropivacaine (Experimental): Ultrasound guided TAP blocks will be performed once patient is in the recovery area. Patients will be placed on their back with their hands resting comfortably above their head. Using an ultrasound guided technique, the ultrasound probe will be positioned on abdominal until the three lateral abdominal wall muscles and TAP are clearly imaged. A two or four inch, 20 gauge needle will be advanced using an in-plane technique. After visual confirmation that the needle tip is in the TAP, 1 ml of preservative free 0.9% sodium chloride will be injected to reconfirm correct placement in the TAP. Then 20 ml of 0.5% ropivacaine will be injected. The procedure will be repeated on the other side.
  Interventions: Drug: 0.5% ropivacaine
- 20 ml per side of 0.9% sodium chloride (Placebo Comparator): Ultrasound guided TAP blocks will be performed once patient is in the recovery area. Patients will be placed on their back with their hands resting comfortably above their head. Using an ultrasound guided technique, the ultrasound probe will be positioned on abdominal until the three lateral abdominal wall muscles and TAP are clearly imaged. A two or four inch, 20 gauge needle will be advanced using an in-plane technique. After visual confirmation that the needle tip is in the TAP, 1 ml of preservative free 0.9% sodium chloride will be injected to reconfirm correct placement in the TAP. Then 20 ml of 0.9% preservative free sodium chloride will be injected. The procedure will be repeated on the other side.
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: 0.5% ropivacaine — 20ml each side of the hip of 0.5% ropivacaine into the transverse abdominis plane after patient is brought to the recovery area after elective cesarean delivery
  Arms: 20 ml per side of 0.5% ropivacaine
Drug: 0.9% sodium chloride — 20ml each side of the hip of 0.9% sodium chloride into the transverse abdominis plane after patient is brought to the recovery area after elective cesarean delivery
  Arms: 20 ml per side of 0.9% sodium chloride

SUMMARY:
The purpose of this study is to determine if injecting a local anesthetic, or numbing medication, above each hip will decrease the amount of narcotic pain medicine that is typically required by a patient after a cesarean delivery. Ultrasound pictures will be used to guide placement of this injection. Either ropivicaine (a type of numbing medication called a local anesthetic) or a placebo (saline) will be injected. For 24 hours, you will be given a button to press when you have pain. When the button is pressed, you will be given a small amount of pain medication called hydromorphone through your IV. You will also be given a pain medication called ketorolac through your IV every 8 hours for 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* ASA class 1 , 2 or 3
* BMI greater than 30 kg/m2 (as recorded at the patient's last clinic appointment or as measured on the day of delivery)
* Scheduled for cesarean section via Pfannenstiel incision (with or without a tubal ligation)
* 150 cm or taller
* Informed consent obtained

Exclusion Criteria:

* ASA class 4
* Age under 18
* Relevant drug allergy
* Contraindication to spinal anesthesia
* Height < 150 cm
* Patient receiving medical therapies considered to result in a tolerance to opioids
* Any other major surgical procedure performed other than cesarean delivery with or without tubal ligation
* Patient with relevant contraindications to ketorolac, such as history of gastrointestinal bleeding or impaired renal function
* Patient refusal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
hydromorphone consumed by patient controlled analgesia in the first 24 hours after cesarean delivery | 24 hours

SECONDARY OUTCOMES:
Categorical pain scores and Visual Analog Scale (VAS) pain scores (at rest and with movement), nausea and sedation will be assessed to evaluate narcotic side effects | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Hart, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Saravanakumar K, Rao SG, Cooper GM. Obesity and obstetric anaesthesia. Anaesthesia. 2006 Jan;61(1):36-48. doi: 10.1111/j.1365-2044.2005.04433.x. PMID 16409341
- [Background] American Society of Anesthesiologists Task Force on Obstetric Anesthesia. Practice guidelines for obstetric anesthesia: an updated report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia. Anesthesiology. 2007 Apr;106(4):843-63. doi: 10.1097/01.anes.0000264744.63275.10. No abstract available. PMID 17413923
- [Result] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577
- [Result] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Result] Belavy D, Cowlishaw PJ, Howes M, Phillips F. Ultrasound-guided transversus abdominis plane block for analgesia after Caesarean delivery. Br J Anaesth. 2009 Nov;103(5):726-30. doi: 10.1093/bja/aep235. Epub 2009 Aug 22. PMID 19700776
- [Result] Tran TM, Ivanusic JJ, Hebbard P, Barrington MJ. Determination of spread of injectate after ultrasound-guided transversus abdominis plane block: a cadaveric study. Br J Anaesth. 2009 Jan;102(1):123-7. doi: 10.1093/bja/aen344. PMID 19059922
- [Result] El-Dawlatly AA, Turkistani A, Kettner SC, Machata AM, Delvi MB, Thallaj A, Kapral S, Marhofer P. Ultrasound-guided transversus abdominis plane block: description of a new technique and comparison with conventional systemic analgesia during laparoscopic cholecystectomy. Br J Anaesth. 2009 Jun;102(6):763-7. doi: 10.1093/bja/aep067. Epub 2009 Apr 17. PMID 19376789